CLINICAL TRIAL: NCT04140097
Title: Predictors of Acute Exacerbation in Patients With COPD - an Observational Study (PACE Trial)
Brief Title: Predictors of Acute Exacerbation in Patients With COPD - an Observational Study
Acronym: PACE
Status: Active, not recruiting | Type: Observational
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Collaborators: GlaxoSmithKline GmbH & Co. KG (Munich, Germany) (Unknown); Coordinating Center for Clinical Trials (KKS; Philipps-University of Marburg, Germany) (Unknown); Research Office (Biostatistics), Paracelsus Medical University (Salzburg, Austria) (Unknown); Fraunhofer ITEM, Biomedical Research in Endstage and Obstructive Lung Disease Hannover (BREATH), German Center for Lung Research (Hannover, Germany) (Unknown); Institute of Laboratory Medicine and Pathobiochemistry, Molecular Diagnostics, Philipps University Marburg (Marburg, Germany) (Unknown)
Responsible Party: Principal Investigator, Klaus Kenn, Professor, Schön Klinik Berchtesgadener Land
Other Study IDs: PACE Trial
Record Dates: First submitted 2019-09-26; First posted 2019-10-25 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD; COPD Exacerbation; COPD Exacerbation Acute
Keywords: Predictor; Development; Pulmonary Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD patients with acute exacerbation
  Interventions: Other: Prospective monitoring of a large variety of parameters
- COPD patients without acute exacerbation
  Interventions: Other: Prospective monitoring of a large variety of parameters

INTERVENTIONS:
Other: Prospective monitoring of a large variety of parameters — Patients will be recruited during an inpatient pulmonary rehabilitation program. This setting offers a unique opportunity to study the phenomenon of an acute exacerbation of the Chronic Obstructive Pulmonary Disease prior to the first visible clinical sign and further on to have a follow up of the underlying mechanisms. All COPD patients that are referred to the reference center for a rehabilitation program will be included after providing written informed consent. Prospectively, a wide range of measurements will be collected. If a patient develops an acute exacerbation there will be a comprehensive diagnostic assessment to differentiate between pulmonary, cardiac or cardio-pulmonary reasons for the exacerbation. The clinical diagnosis of an AECOPD will be made by a pulmonologist according to criteria of international guidelines within the first 24h of clinical symptoms suggestive of an exacerbation.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a lung disease characterized by respiratory problems and poor airflow with dyspnea and cough being the main symptoms. Acute exacerbations of COPD (AECOPD) are the most important events for patients with COPD that have a negative impact on patients´ quality of life, accelerate disease progression, and can result in hospital admissions and death. It is of major clinical importance to determine predictors of an AECOPD and to identify patients who are at high risk for developing an acute exacerbation and/or to detect the beginning of or prevent an ongoing acute exacerbation as early as possible. Until now, research in the field of AECOPD has gathered and analyzed data only after manifestation of AECOPD until recovery and most of them used a retrospective study design. Therefore, the aim of this prospective trial is to collect clinical data in patients prior to the first visible clinical signs of an AECOPD to investigate potential early predictors of an AECOPD.

DETAILED DESCRIPTION:
In total, 355 COPD patients will be included prospectively to this study during a 3-week inpatient pulmonary rehabilitation programme at the Schoen Klinik Berchtesgadener Land, Schoenau am Koenigssee, (Germany). All patients will be closely monitored from admission to the study. Measures of lung function, blood samples, breath sampling, exercise tests, physical activity monitoring, cardiac parameters, quality of life and a symptom diary will be recorded regularly. Prior knowledge from this programme suggest that about 15% of patients will develop an AECOPD during this observational phase. If a patient develops an AECOPD there will be a comprehensive diagnostic assessment to differentiate between cardiac, pulmonary or cardio-pulmonary reasons for the AECOPD and to identify the type of exacerbation. The clinical diagnosis and management of an AECOPD will be determined by a pulmonologist according to criteria of international guidelines within the first 24h after the onset of clinical symptoms suggestive of an exacerbation. Collected clinical data from the days prior to AECOPD will be analyzed comprehensively to identify parameters with high prediction power for AECOPD. Furthermore, patients will perform follow-up measures at 6, 12 and 24 months following the initial observational phase (PR phase).

A wide range of predictor screening methods will be applied to identify significant predictors including cross tabulation tables, correlations, generalized linear models, mixed models, generalized estimation equation models and various predictor screening methods based on variable selection algorithms.

Study objectives Primary endpoint: To prospectively identify potential early, respiratory and/ or cardiac clinical predictors, laboratory parameters, breath print analyses and/ or changes in lung function and physical activity prior to an AECOPD in COPD patients.

Secondary endpoint(s):

1. To identify potential mechanisms explaining the nature and composition of an acute exacerbation in COPD patients
2. To identify and differentiate patterns of acute COPD exacerbation versus cardiac failure in COPD patients
3. To investigate the potential role of an electronic-nose to capture exhaled breath metabolomic profiles for the early detection of an acute exacerbation in COPD patients ("COPD pre exacerbation breath print")
4. To identify parameters influencing mortality and other adverse events in the total study cohort at 6, 12 and 24 months follow up

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of Chronic Obstructive Pulmonary Disease according to Global Association for Obstructive Lung Disease stage II to IV
* the ability to follow the rehabilitation protocol
* provided written informed consent

Exclusion Criteria:

- current primary diagnosis of asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic Obstructive Pulmonary Disease that are referred to an inpatient pulmonary rehabilitation program at the reference center.
Sampling Method: Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline laboratory parameters at day 21 | baseline and day 21
  following Parameters will be collected: c-reactive protein, cardiac Troponin I, hemoglobin A1c, Interleukin-1 beta, Interleukin-2, Interleukin-6, Interleukin 8, N-terminal probrain natriuretic peptide, Tumor necrosis factor alpha
Change from day 1 of an acute exacerbation in laboratory parameters at day 5 | day 1 and 5 in case of an acute exacerbation
  following Parameters will be collected: c-reactive protein, cardiac Troponin I, hemoglobin A1c, Interleukin-1 beta, Interleukin-2, Interleukin-6, Interleukin 8, N-terminal probrain natriuretic peptide, Tumor necrosis factor alpha
Change from baseline lung function at day 21 | baseline and day 21
  following Parameters will be collected: forced expiratory volume in 1 sec, forced vital capacity, total lung capacity, residual volume
Change from day 1 of an acute exacerbation in lung function at day 5 | day 1 and 5 in case of an acute exacerbation
  following Parameters will be collected: forced expiratory volume in 1 sec, forced vital capacity, total lung capacity, residual volume
Change from baseline Cardiac Doppler echocardiography at day 21 | baseline and day 21
  Left and right heart echocardiography will be performed
Change from day 1 of an acute exacerbation in Cardiac Doppler echocardiography at day 5 | day 1 and 5 in case of an acute exacerbation
  Left and right heart echocardiography will be performed
Change from baseline breath volatile organic compounds Analysis to day 4, 8, 11, 15 and 18 | day 1, 4, 8, 11, 15, 18
  breath samples will be analyzed by ion-mobility spectrometry and gaschromatography/mass spectrometry
Change in baseline exercise Performance at day 21 | day 1 and 21
  following tests will be performed: 6-Minute walk test, sit-to-stand-test, Peak quadriceps and Hand grip force,
Change from baseline Quality of life assessed by Short Form - 36 Questionnaire at days 21, day 180, day360, day 720 | baseline, day 21, day 180, day 360, day 720
  the scale of the physical and mental Health component summary score ranges from 0 to 100 Points with higher scores indicating better Quality of lif
Change from baseline functional status assessed by Modified Medical Research Counsil score at days 21, day 180, day360, day 720 | baseline, day 21, day 180, day 360, day 720
  the score ranges from category 0 to 4 with higher scores indicating higher impairment in function status
Change from baseline anxiety status assessed by Chronic Obstructive Pulmonary Disease Anxiety Questionnaire at days 21, day 180, day360, day 720 | baseline, day 21, day 180, day 360, day 720
  the total score ranges from 0 to 112 Points with higher scores indicating worse anxiety status
Change from baseline Depression status assessed by Patient Health Questionnaire 9 at days 21, day 180, day360, day 720 | baseline, day 21, day 180, day 360, day 720
  the total score ranges from 0 to 27 Points with higher scores indicating worse Depression symptoms
Change from baseline disease specific Quality of life assessed by Chronic Obstructive Pulmonary Disease Assessment Test at days 21, day 180, day360, day 720 | baseline, (day 1 and 5 in case of an acute exacerbation), day 21, day 180, day 360, day 720
  total score ranges from 0 to 40 points with higher scores indicating worse quality of life
Self-reported patient diary | once daily from day 1 to day 21
  The EXAcerbations of Chronic pulmonary disease Tool will be used
physical activity monitoring | continuous monitoring from day 1 to day 21
  Using the Actigraph device following Parameters will be collected: steps per day and physical activity levels
Change in Survival Status from baseline at 6, 12 and 24 months | baseline, at 6, 12 and 24 months
  Survival Status will be assessed by phone calls
cough events | Recording from day 1 to day 21 at night only
  Number of nocturnal cough events recorded by NELA sound device (Carepath)
Self-reported patient symptom diary | Once daily from day 1 to day 21
  The COPD Exacerbation Recognition Tool (CERT) is used. The CERT asks about symptoms of increased cough, sputum production, shortness of breath, labored breathing, and reduced physical activity. The total score ranges from 0 (symptoms as usual) to 5 (severe deterioration compared to usual).

CONTACTS AND LOCATIONS:
Locations (1):
- Schoen Klinik Berchtesgadener Land, Schönau am Königssee, Germany

REFERENCES:
- [Derived] Gloeckl R, Jones PW, Kroll D, Jarosch I, Schneeberger T, Claussen J, Schmidt P, Vogelmeier CF, Kenn K, Koczulla AR. Can Patient Education Lead the Way? Head-To-Head Comparison of EXACT and CERT for Early Recognition of Acute COPD Exacerbations. Respirology. 2025 Nov 30. doi: 10.1002/resp.70170. Online ahead of print. PMID 41320645
- [Derived] Kenn K, Gloeckl R, Leitl D, Schneeberger T, Jarosch I, Hitzl W, Alter P, Sczepanski B, Winterkamp S, Boensch M, Schade-Brittinger C, Skevaki C, Holz O, Jones PW, Vogelmeier CF, Koczulla AR. Protocol for an observational study to identify potential predictors of an acute exacerbation in patients with chronic obstructive pulmonary disease (the PACE Study). BMJ Open. 2021 Feb 8;11(2):e043014. doi: 10.1136/bmjopen-2020-043014. PMID 33558356